CLINICAL TRIAL: NCT01754636
Title: Elderly Patients With Colorectal Cancer in Clinical Trials: Factors Associated With Non Inclusion
Brief Title: Inclusion of Elderly Patients With Colorectal Cancer in Clinical Trials
Acronym: SAGE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 11006
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal neoplasms; Elderly; Randomized clinical trials; Inclusion.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elderly patients: patients aged 65 years old or older : no intervention
  Interventions: Other: No intervention
- "Young" patients: patients aged 18-64 years (added by amendment n°3 -02/2014) : no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Background: Inadequate representation of elderly cancer patients in randomized clinical trials (RCTs) leading to a lack of external validity thereby an uncertainty regarding benefit-risk balance of cancer treatment in elderly, especially chemotherapy.

Hypothesis: The eligibility criteria explain only a part of the under-representation of elderly patients in trials. We make the assumptions that 1) Among the eligible, the invitation to participate in a trial and inclusion are inversely related to age, 2) Among the eligible, there are patients, practitioner, or organization factors that would explain the non inclusion of elderly patients.

Objectives:

1) To assess, in elderly patients with colorectal cancer, the proportions of patients:

1. eligible at least to one RCT
2. invited to participate
3. included 2)

a) Compare proportions among elderly patients to those of the comparator group of "young" subjects (age ≥ 18 and <65 years) (added by amendment n°3 accepted 18/02/2014) b)To identify factors associated with the non-invitation and the non-inclusion in RCT.

Material and methods:

Study design: A multicentric prospective cohort survey Population: all patients aged 18 years or more (added by amendment n°3 - 02/2014) with a colorectal cancer followed in one of the participating centers.

Data collection:

* At baseline: Patient characteristics (including SOCIO-demographic, oncologic and geriatric data) will be collected. Organization factors (e.g. clinical research team) will be collected.
* Follow-up: the patient will be followed for potential invitation and inclusion in one RCT. Reasons of non-invitation or non-inclusion will be assessed.

Number of subjects needed: 696 (553 elderly patients and 143 "young" patients) Number of centers : 7 (added by amendment n°3 - 02/2014)

Ethical aspects: each patient will give his oral informed consent. The International Review Board of Mondor Hospital (CPP Ile-de-France IX) gave its approval in December 2012.

ELIGIBILITY:
Inclusion Criteria:

Patient aged of of 18 years and older (modified by amendment n°3 - 02/2014)

For a diagnosed colorectal cancer (CRC) irrespective of the stage

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population: all patients aged 18 years or more with a colorectal cancer followed in one of the participating centers (amendment n°3 - 02/2014)
Sampling Method: Non-Probability Sample
Enrollment: 707 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Inclusion in at least one Clinical trial (amendment n°3 -02/2014) | At the end of recruiting period (nov. 2012 - nov. 2016)

SECONDARY OUTCOMES:
Eligibility to participate in in at least one Clinical trial (amendment n°3 -02/2014) | Four years
Invitation to participate in in at least one Clinical trial (amendment n°3 -02/2014) | Four years

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, Val de Marne, France

REFERENCES:
- [Background] Aparicio T, Navazesh A, Boutron I, Bouarioua N, Chosidow D, Mion M, Choudat L, Sobhani I, Mentre F, Soule JC. Half of elderly patients routinely treated for colorectal cancer receive a sub-standard treatment. Crit Rev Oncol Hematol. 2009 Sep;71(3):249-57. doi: 10.1016/j.critrevonc.2008.11.006. Epub 2009 Jan 7. PMID 19131256
- [Background] Lewis JH, Kilgore ML, Goldman DP, Trimble EL, Kaplan R, Montello MJ, Housman MG, Escarce JJ. Participation of patients 65 years of age or older in cancer clinical trials. J Clin Oncol. 2003 Apr 1;21(7):1383-9. doi: 10.1200/JCO.2003.08.010. PMID 12663731
- [Derived] Canoui-Poitrine F, Lievre A, Dayde F, Lopez-Trabada-Ataz D, Baumgaertner I, Dubreuil O, Brunetti F, Coriat R, Maley K, Pernot S, Tournigand C, Hagege M, Aparicio T, Paillaud E, Bastuji-Garin S. Inclusion of Older Patients with Cancer in Clinical Trials: The SAGE Prospective Multicenter Cohort Survey. Oncologist. 2019 Dec;24(12):e1351-e1359. doi: 10.1634/theoncologist.2019-0166. Epub 2019 Jul 19. PMID 31324663